CLINICAL TRIAL: NCT01869335
Title: A Randomized Study Comparing ex Vivo MRI Versus Radiography of Breast Specimens in Evaluating Tumor-free Margins After Surgical Resection of Breast Microcalcifications
Brief Title: A Study Comparing ex Vivo MRI Versus Radiography of Breast Specimens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Roberto Agresti, MD, MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/13
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; MRI; mammography; microcalcifications; Local staging of breast microcalcifications; Evaluation of ex vivo MRI for breast malignancies detected by MRI only
MeSH Terms: conditions — Breast Neoplasms; Calcinosis | interventions — Radiography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- radiography (Active Comparator): Arm1: patients undergo mammographic localizations and radiography of the specimen after surgical resection.
  Interventions: Device: radiography
- MRI (magnetic resonance imaging) (Active Comparator): Arm2: patients undergo MRI localization and ex vivo MRI after surgical resection.
  Interventions: Device: MRI (magnetic resonance imaging)

INTERVENTIONS:
Device: radiography
  Arms: radiography
Device: MRI (magnetic resonance imaging)
  Arms: MRI (magnetic resonance imaging)

SUMMARY:
Radiography of breast specimens is currently the only radiological procedure used to verify removal of microcalcifications and presence of tumor-free margins after breast surgical resection. Ex vivo MRI will be tested for its ability to detect residual tumor tissue not detected by radiography in resected breast tumor specimens and/or its ability to verify tumor-free margins in breast cancer detected by MRI only.

ELIGIBILITY:
Inclusion Criteria:

* Women with malignant breast disease identified by microcalcifications without clinically evident disease
* Women candidate to breast preserving surgery

Exclusion Criteria:

* Cardiac pacemaker, defibrillators, cardiac monitors
* Brain stimulators, implantable spinal stimulators
* Vascular and aneurismal clips
* Hemostatic clips
* Infusion pumps
* Glaucoma drainage implants
* Metallic foreign body positioned in vital organ of the patients
* Some heart valves
* Some vascular access ports, infusion pumps and catheters
* Permanent contraceptive tubal device
* Kidney disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of Magnetic Resonance Imaging (MRI) versus radiography in evaluating tumor-free margins in breast cancer specimens | 2 years
  Diagnostic efficacy will be evaluated by statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Background] Elshof LE, Rutgers EJ, Deurloo EE, Loo CE, Wesseling J, Pengel KE, Gilhuijs KG. A practical approach to manage additional lesions at preoperative breast MRI in patients eligible for breast conserving therapy: results. Breast Cancer Res Treat. 2010 Dec;124(3):707-15. doi: 10.1007/s10549-010-1064-z. Epub 2010 Jul 22. PMID 20652399